CLINICAL TRIAL: NCT01654315
Title: Robotic Brace Incorporating EMG for Moderate Affected Arm Impairment After Stroke
Brief Title: Robotic Brace Incorporating Electromyography for Moderate Affected Arm Impairment After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011H0215
Record Dates: First submitted 2012-05-16; First posted 2012-07-31 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Hemiparesis
Keywords: RTP Only Group; Myomo Only Group; Myomo + RTP Group
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: Myomo Only Group (Experimental): Experimental: Myomo Only Group Patients are administered rehabilitative therapy known as "repetitive task specific practice" (RTP) using only the Myomo robotic device targeting their affected arms on 3 days/week, in 1/2 hour increments, during an 8-week period.
  Interventions: Device: Myomo Robotic Arm
- Experimental: Myomo + RTP Group (Experimental): Experimental: Myomo + RTP Group Patients are administered rehabilitative therapy using both the Myomo robotic device and RTP targeting their affected arms on 3 days/week in 1/2 hour increments, during an 8 week period. These patients engage in activities that emphasize use of their affected arms repetitively, with the device providing assistance as needed with movement through the arm's range of motion. As patients progress, the amount of assistance provided by the device during the activities is reduced.
  Interventions: Device: Myomo Robotic Arm
- Active Comparator: RTP Group (Active Comparator): Active Comparator: RTP Group Patients are administered rehabilitative therapy using only RTP that is targeting their affected arms on 3 days/week during a 8 week period. In this condition, patients engage in activities that emphasize use of their affected arms repetitively, with the therapist providing assistance as needed with movement through the arm's range of motion. As patients progress, the amount of assistance provided by the therapist during the activities is reduced.
  Interventions: Behavioral: RTP Standard Therapy

INTERVENTIONS:
Device: Myomo Robotic Arm — Patients are administered rehabilitative therapy (repetitive task specific therapy,, also known as "RTP' in this study) using only the Myomo robotic device targeting their affected arms on 3 days/week during a 8 week period. These patients engage in RTP, which consists of a battery of activities that emphasize use of their affected arms repetitively, with the device providing assistance as needed with movement through the arm's range of motion.
  Arms: Experimental: Myomo + RTP Group; Experimental: Myomo Only Group
Behavioral: RTP Standard Therapy — Active Comparator: RTP Group Patients are administered rehabilitative therapy using only RTP that is targeting their affected arms on 3 days/week during a 8 week period. In this condition, patients engage in activities that emphasize use of their affected arms repetitively, with the therapist providing assistance as needed with movement through the arm's range of motion. As patients progress, the amount of assistance provided by the therapist during the activities is reduced.
  Arms: Active Comparator: RTP Group

SUMMARY:
Of the 5.7 million stroke survivors in the United States, up to 80% exhibit significant weakness in one arm (called "hemiparesis"). This devastating impairment undermines performance of valued activities and quality of life. Although rehabilitation is commonly provided, conventional affected arm rehabilitative strategies have negative evidence, or no evidence, supporting their use. Thus, there remains a need for evidence-based rehabilitative strategies for arm hemiparesis.

Newer rehabilitative approaches emphasize repetitive, task-specific practice (RTP) incorporating the affected arm. However, many of these promising regimens require participation in intensive therapies, and most are only efficacious on the least impaired patients. Thus, there remains a need for an efficacious, practical RTP technique to address moderate affected arm hemiparesis.

To address the above shortfalls, one of the investigators team members piloted an innovative brace integrating electromyography (EMG) and robotics. In his case series, 8 stroke patients exhibiting moderate arm impairment successfully participated in RTP, with the brace (called the "Myomo") detecting and augmenting their movement attempts. Aided by the Myomo, participation in the RTP regimen reduced subjects' affected arm impairment and spasticity. The next logical step is to test Myomo + RTP efficacy using randomized controlled methods and an appropriate sample size.

DETAILED DESCRIPTION:
The primary objective of this small efficacy study is to collect randomized, controlled pilot data estimating clinical effectiveness of this combined, EMG/robotics approach in conjunction with RTP. A unique adjunct will be acquisition of biomechanical data as an outcome measure. Based on pilot data, the central hypothesis is that Myomo therapy with RTP will exhibit significant impairment reductions. We will test the central hypothesis and accomplish the objective by pursuing the following specific aims:

Specific Aim 1: Compare efficacy of Myomo + RTP with RTP only and Myomo only on affected arm impairment. Thirty stroke patients exhibiting moderate affected arm deficits will be randomly assigned to receive: (a) Myomo combined with RTP (Myomo + RTP); (b) RTP only (RTP), which constitutes the most frequently used regimen in clinical environments;2,3 or (c) Myomo therapy only (Myomo). The current study design will determine the additive effect of Myomo training to RTP, while also discerning the relative efficacy of RTP only or Myomo use only. The intended duration of contact will be equivalent across groups.

Affected arm impairment, the primary study outcome, will be measured by the upper extremity section of the Fugl-Meyer Impairment Scale (FM), the primary outcome measure. The FM will be administered by a blinded rater twice before intervention, immediately post-intervention (POST), and two months post-intervention (POST-2) with POST serving as the primary study endpoint. The primary study hypothesis is that subjects in the Myomo + RTP group will exhibit significantly larger FM score changes than Myomo or RTP subjects at POST. It is also hypothesized that these changes will be sustained at POST-2.

Specific Aim 2: Determine the impact of Myomo + RTP on affected arm outcomes. The investigators will administer the Arm Motor Ability Test (AMAT), to all subjects before intervention, at POST, and at POST-2. When compared to their scores before intervention, it is hypothesized that Myomo + RTP subjects will exhibit significantly larger AMAT score changes,than subjects in the other groups at POST. These differences will be sustained at POST-2.

ELIGIBILITY:
Inclusion Criteria:

* upper extremity Fugl Meyer score >10-< 25 (i.e., subject must score between (and including) 10 and 25 on the UE FM at the baseline screening appointment only)
* presence of volitionally activated EMG signal from the paretic biceps brachii of at least 5 ųV in amplitude
* stroke experienced > 1 month prior to study enrollment
* a score > 24 on the Folstein Mini Mental Status Examination (MMSE)
* age > 35 < 85
* have experienced one stroke
* discharged from all forms of physical rehabilitation
* Myomo brace fits on affected arm properly and without discomfort (i.e., no red marks or discomfort observed in 10 minutes of use during fitting).
* < 35 years old
* excessive pain in the affected hand, arm or shoulder, as measured by a score > 5 on a 10-point visual analog scale
* excessive spasticity at the affected elbow, as defined as a score of > 4 on the Modified Ashworth Spasticity Scale
* currently participating in any experimental rehabilitation or drug studies
* apraxia (< 2.5 on the Alexander scale)
* severe sensory loss in affected hand (Nottingham sensory scale at least 75% of normal)
* severe language deficits (score < 2 on NIH Stroke Scale question 9)
* Stroke that occurred in the brainstem (corticospinal tracts are the final pathway for the motor system, and are frequently damaged in brainstem strokes. These individuals are hypothesized to be less likely to benefit from the cortical plasticity seen with exercise therapy, and are therefore excluded from this study.)
* A current medical history of uncontrolled cardiovascular, or pulmonary disease, or other disease that would preclude involvement in a therapeutic treatment (Subjects must be able to tolerate a one-hour upper-extremity therapy session.)
* History of neurological disorder other than stroke (other neurological disorders may affect the upper extremity motor performance of subjects.); (11) Other significant pain or skin irritation in the upper extremity that would be exacerbated if by the use of the brace (While wearing the brace, the system is pressed close to the upper arm and strapped around it. (If the subject suffers from dermal breakdown or other skin conditions that may be aggravated by such a situation, they should not be involved in the study.)
* Substantial contracture of elbow, defined as > 20 degrees of elbow flexion, as measured at the baseline evaluation. (The system cannot work in the presence of reduced range of motion due to contractures.).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Page, PhD,M.S., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Myomo Only Group: Experimental: Myomo Only Group Patients are administered rehabilitative therapy using only the Myomo robotic device targeting their affected arms on 3 days/week during a 8 week period.
  Myomo Robotic Arm: Patients are administered rehabilitative therapy using only the Myomo robotic device targeting their affected arms on 3 days/week during a 8 week period.
- Experimental: Myomo + RTP Group: Experimental: Myomo + RTP Group Patients are administered rehabilitative therapy using both the Myomo robotic device and RTP targeting their affected arms on 3 days/week during a 8 week period.
  Myomo Robotic Arm: Patients are administered rehabilitative therapy using only the Myomo robotic device targeting their affected arms on 3 days/week during a 8 week period.
- Active Comparator: RTP Group: Active Comparator: RTP Group Patients are administered rehabilitative therapy using only RTP that is targeting their affected arms on 3 days/week during a 8 week period.
  Myomo Robotic Arm: Patients are administered rehabilitative therapy using only the Myomo robotic device targeting their affected arms on 3 days/week during a 8 week period.
Period: Overall Study
Arm/Group | Experimental: Myomo Only Group | Experimental: Myomo + RTP Group | Active Comparator: RTP Group
Started | 15 | 10 | 9
Completed | 15 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Myomo Only Group | Experimental: Myomo + RTP Group | Active Comparator: RTP Group | Total
Number analyzed (Participants) | 15 | 10 | 9 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.69 (8.6) | 52.28 (13.0) | 57.22 (7.7) | 54.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 11
  Male | 10 | 7 | 6 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 10 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Impairment in the Affected Upper Extremity as Measured by the Fugl Meyer Scale.
Description: The upper extremity section of the Fugl-Meyer Scale (FM) will assess whether changes occur in paretic upper extremity motor impairment. The FM has been used extensively in stroke recovery studies, and is highly recommended for "use in clinical trials designed to evaluate changes in motor impairment following stroke." The items on the measure require the subject to perform various movements with the affected upper extremity, and each item is scored from 0 (cannot perform) to 2 (performs normally). Item are then summed for a total score. The total score ranges are 0 to 66, with a higher score representing less upper extremity impairment (and, thus, a relatively "better" score on the measure than a lower score).
Time Frame: Administered twice before the intervention period. These two scores are averaged to provide a composite score that is compared to average score for each group that is collected 1 week after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: Myomo Only Group | Experimental: Myomo + RTP Group | Active Comparator: RTP Group
Number analyzed (Participants) | 15 | 10 | 9
units on a scale | 19.6 (3.8) | 18.0 (5.9) | 17.6 (4.4)

2. Secondary Outcome: Arm Motor Ability Test (AMAT)
Description: The Arm Motor Activity Test (AMAT) was the secondary outcome for this study and was used to determine whether changes occur in activity limitation. The AMAT is a 13-item test in which valued activities are rated according to a functional ability scale that examines affected limb use 0 = no use, 1 = very slight use, 2 = slight use, 3 = moderate use, 4 = almost normal use, 5 = normal use;) and a Quality of Movement Scale (0 = no use, 1 = very poor, 2 = poor, 3 = fair, 4 = almost normal, 5 = normal. ). Therefore, the highest score that one can attain on either scale is 65.0 (which would mean that the person scored a perfect score of "5" on each of the thirteen items).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: Myomo Only Group | Experimental: Myomo + RTP Group | Active Comparator: RTP Group
Number analyzed (Participants) | 15 | 10 | 9
units on a scale | 29.21 (8.67) | 28.62 (8.38) | 25.33 (5.24)

ADVERSE EVENTS:
Arm/Group | Experimental: Myomo Only Group | Experimental: Myomo + RTP Group | Active Comparator: RTP Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No